CLINICAL TRIAL: NCT04234113
Title: A Multicenter Open-label Phase 1/1b Study to Evaluate the Safety and Preliminary Efficacy of SO-C101 as Monotherapy and in Combination With Pembrolizumab in Patients With Selected Advanced/Metastatic Solid Tumors
Brief Title: Study of Nanrilkefusp Alfa Alone and With Pembrolizumab in Adult Patients With Advanced/Metastatic Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to lack of efficacy shown at the time of the interim analysis.
Sponsor: SOTIO Biotech AG (Industry)
Collaborators: SOTIO Biotech a.s. (Industry)
Responsible Party: Sponsor
Organization: Sotio Biotech Inc. (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SC103; AURELIO-03 (Other: SOTIO Biotech AG); 2018-004334-15 (EudraCT Number)
Record Dates: First submitted 2019-11-14; First posted 2020-01-21 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2024-09

CONDITIONS: Thyroid Cancer; Renal Cell Carcinoma; Non Small Cell Lung Cancer; Small-cell Lung Cancer; Bladder Cancer; Melanoma; Merkel Cell Carcinoma; Skin Squamous Cell Carcinoma; Microsatellite Instability High; Triple Negative Breast Cancer; Mesothelioma; Thymic Cancer; Cervical Cancer; Biliary Tract Cancer; Hepatocellular Carcinoma; Ovarian Cancer; Gastric Cancer; Head and Neck Squamous Cell Carcinoma; Anal Cancer
Keywords: Thyroid Cancer; Renal Cell Carcinoma; Non Small Cell Lung Cancer; Small-cell Lung Cancer; Bladder Cancer; Melanoma; Merkel Cell Carcinoma; Skin Squamous Cell Carcinoma; Microsatellite Instability High; Triple Negative Breast Cancer; Mesothelioma; Thymic Cancer; Cervical Cancer; Biliary Tract Cancer; Hepatocellular Carcinoma; Ovarian Cancer; Gastric Cancer; Head and Neck Squamous Cell Carcinoma; Anal Cancer
MeSH Terms: conditions — Thyroid Neoplasms; Carcinoma, Renal Cell; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Urinary Bladder Neoplasms; Melanoma; Carcinoma, Merkel Cell; Triple Negative Breast Neoplasms; Mesothelioma; Thymus Neoplasms; Uterine Cervical Neoplasms; Biliary Tract Neoplasms; Carcinoma, Hepatocellular; Ovarian Neoplasms; Stomach Neoplasms; Squamous Cell Carcinoma of Head and Neck; Anus Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Experimental: Part A (nanrilkefusp alfa monotherapy) (Experimental): Drug: Nanrilkefusp alfa
  Interventions: Drug: Nanrilkefusp alfa
- Experimental: Part B (nanrilkefusp alfa combined with pembrolizumab) (Experimental): Drug: Nanrilkefusp alfa Drug: Pembrolizumab
  Interventions: Drug: Nanrilkefusp alfa; Drug: Pembrolizumab
- Experimental: Part A1 (nanrilkefusp alfa divided dosing, monotherapy) (Experimental): Drug: Nanrilkefusp alfa, twice a day as 2 divided doses (50%:50%)
  Interventions: Drug: Nanrilkefusp alfa
- Experimental: Part B1 (nanrilkefusp alfa divided dosing, combined with pembrolizumab) (Experimental): Drug: Nanrilkefusp alfa, twice a day as 2 divided doses (50%:50%) Drug: Pembrolizumab
  Interventions: Drug: Nanrilkefusp alfa; Drug: Pembrolizumab
- Experimental: Part D (nanrilkefusp alfa monotherapy, expansion at the RP2D identified in Part A) (Experimental): Drug: Nanrilkefusp alfa Indications: Relapsed/refractory advanced/metastatic renal cell carcinoma, relapsed/refractory advanced/metastatic skin squamous-cell carcinoma, relapsed/refractory advanced/metastatic melanoma
  Interventions: Drug: Nanrilkefusp alfa
- Part D1 (nanrilkefusp alfa divided dosing, monotherapy, expansion at the RP2D identified in Part A1) (Experimental): Drug: Nanrilkefusp alfa, twice a day as 2 divided doses (50%:50%) Indications: Relapsed/refractory advanced/metastatic renal cell carcinoma, relapsed/refractory advanced/metastatic skin squamous-cell carcinoma, relapsed/refractory advanced/metastatic melanoma
  Interventions: Drug: Nanrilkefusp alfa

INTERVENTIONS:
Drug: Nanrilkefusp alfa — A fusion protein which consists of the N-terminal sushi domain of human IL-15 receptor α covalently coupled via a linker of 20 amino acids to human IL-15
  Other Names: SOT101; SO-C101; RLI-15
Drug: Pembrolizumab — A humanized IgG4 monoclonal antibody with high specificity of binding to the PD-1 receptor
  Other Names: KEYTRUDA®
  Arms: Experimental: Part B (nanrilkefusp alfa combined with pembrolizumab); Experimental: Part B1 (nanrilkefusp alfa divided dosing, combined with pembrolizumab)

SUMMARY:
A multicenter open-label phase 1/1b study to evaluate the safety and preliminary efficacy of nanrilkefusp alfa as monotherapy and in combination with pembrolizumab in patients with selected advanced/metastatic solid tumors

DETAILED DESCRIPTION:
This study will assess the safety and tolerability of nanrilkefusp alfa administered as monotherapy and in combination with an anti-PD-1 antibody (pembrolizumab) in patients with selected relapsed/refractory advanced/metastatic solid tumors (renal cell carcinoma, non-small cell lung cancer, small-cell lung cancer, bladder cancer, melanoma, Merkel-cell carcinoma, skin squamous-cell carcinoma, microsatellite instability high solid tumors, triple-negative breast cancer, mesothelioma, thyroid cancer, thymic cancer, cervical cancer, biliary tract cancer, hepatocellular carcinoma, ovarian cancer, gastric cancer, head and neck squamous-cell carcinoma, and anal cancer).

ELIGIBILITY:
Inclusion criteria:

* Patients with selected histologically or cytologically confirmed advanced and/or metastatic solid tumors who are refractory to or intolerant of existing therapies known to provide clinical benefit for their condition.
* ECOG performance score 0-1. Patients with ECOG performance score 2 to be discussed with the sponsor's medical monitor to be agreed for inclusion.
* Estimated life expectancy of ≥3 months
* Washout periods: 4 weeks for chemotherapy, 4 weeks or 5 half-lives (whichever shorter) for biologic agents including immuno-oncology therapy and 4 weeks from major surgeries, definitive radiotherapy and 2 weeks after palliative radiotherapy
* At least one measurable lesion per iRECIST in a non-irradiated port. If in a previously irradiated port, must have demonstrated progression since best response to radiation therapy.
* Have fully recovered from previous treatment to grade ≤1 toxicity (excluding alopecia) or have stable grade 2 neuropathy
* Adequate organ system function
* Negative serum pregnancy test, if woman of child-bearing potential (non-childbearing is defined as greater than one year postmenopausal or surgically sterilized).
* Accessible tumor tissue available for fresh biopsy

Exclusion criteria:

* Untreated central nervous system metastases and/or leptomeningeal carcinomatosis
* Known additional malignancy that is progressing and/or requires active treatment
* Prior exposure to drugs that are agonists of IL-2- or IL-15-like but not limited to rhIL-15 (NCI), ALT-803 (ALTOR), NKTR-214 (Nektar)
* History of and current interstitial lung disease or fibrosis and pneumonitis; patients with clinically significant or oxygen requiring chronic obstructive pulmonary disease or any chronic inflammatory disease (sarcoidosis etc.)
* Has received a live vaccine within 30 days of planned start of study therapy
* Absolute white blood cell count ≤2.0 ×10e9/L
* Absolute neutrophil count ≤1.0 ×10e9/L
* Platelet count ≤100×10e9/L
* Pregnant or breastfeeding women
* Any active autoimmune disease or a documented history of autoimmune disease, poorly controlled asthma, or history of syndrome that required systemic steroids (except the allowed doses) or immunosuppressive medications, except for patients with vitiligo or resolved childhood asthma/atopy
* Specific co-morbidities
* Parts B and B1:

  * Is hypersensitive to any of the ingredients of pembrolizumab drug product (KEYTRUDA®)
  * History of solid organ transplantation or hematopoietic stem cell transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2019-06-13 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-11-27 (Actual)

PRIMARY OUTCOMES:
Part A: Number of participants with dose-limiting toxicities (DLTs) | Through Cycle 1 (21 days)
  Adverse events (AEs) as per NCI CTCAE version 5.0:
  * Grade 5 not related to disease progression or other causes
  * Grade ≥3 non-hematologic toxicity; exceptions: grade 3 nausea, vomiting or diarrhea controlled in 72 hours; grade 3 fatigue <5 days; grade ≥3 correctable electrolyte abnormalities <72 hours and no clinical complications; grade ≥3 amylase or lipase without clinical pancreatitis
  * Hy's law cases
  * Grade 3 AST or ALT or grade 3 bilirubinemia >5 days
  * Hematologic DLTs:
    * Grade 4 neutropenia or thrombocytopenia >7 days
    * Febrile neutropenia
    * Grade ≥3 thrombocytopenia with bleeding
  * Grade 4 immune-related AEs
  * Grade 3 or 4 non-infectious pneumonitis
  * Grade 3 immune-related AEs, excluding colitis, hepatitis, and pneumonitis, not downgrading to grade ≤2 in 3 days despite maximal supportive care including systemic corticosteroids or to grade 1 or baseline in 14 days
  * Grade 2 pneumonitis not downgrading to grade 1 in 3 days
  * Grade 3 colitis
Part A1: Number of participants with DLTs | Through Cycle 1 (21 days)
  AEs as per NCI CTCAE version 5.0:
  * Grade 5 not related to disease progression or other causes
  * Grade ≥3 non-hematologic toxicity; exceptions: grade 3 nausea, vomiting or diarrhea controlled in 72 hours; grade 3 fatigue <5 days; grade ≥3 correctable electrolyte abnormalities <72 hours and no clinical complications; grade ≥3 amylase or lipase without clinical pancreatitis
  * Hy's law cases
  * Grade 3 AST or ALT or grade 3 bilirubinemia >5 days
  * Hematologic DLTs:
    * Grade 4 neutropenia or thrombocytopenia >7 days
    * Febrile neutropenia
    * Grade ≥3 thrombocytopenia with bleeding
  * Grade 4 immune-related AEs
  * Grade 3 or 4 non-infectious pneumonitis
  * Grade 3 immune-related AEs, excluding colitis, hepatitis, and pneumonitis, not downgrading to grade ≤2 in 3 days despite maximal supportive care including systemic corticosteroids or to grade 1 or baseline in 14 days
  * Grade 2 pneumonitis not downgrading to grade 1 in 3 days
  * Grade 3 colitis
Part B: Number of participants with DLTs | Through Cycle 1 (21 days)
  AEs as per NCI CTCAE version 5.0:
  * Grade 5 not related to disease progression or other causes
  * Grade ≥3 non-hematologic toxicity; exceptions: grade 3 nausea, vomiting or diarrhea controlled in 72 hours; grade 3 fatigue <5 days; grade ≥3 correctable electrolyte abnormalities <72 hours and no clinical complications; grade ≥3 amylase or lipase without clinical pancreatitis
  * Hy's law cases
  * Grade 3 AST or ALT or grade 3 bilirubinemia >5 days
  * Hematologic DLTs:
    * Grade 4 neutropenia or thrombocytopenia >7 days
    * Febrile neutropenia
    * Grade ≥3 thrombocytopenia with bleeding
  * Grade 4 immune-related AEs
  * Grade 3 or 4 non-infectious pneumonitis
  * Grade 3 immune-related AEs, excluding colitis, hepatitis, and pneumonitis, not downgrading to grade ≤2 in 3 days despite maximal supportive care including systemic corticosteroids or to grade 1 or baseline in 14 days
  * Grade 2 pneumonitis not downgrading to grade 1 in 3 days
  * Recurrent grade 2 pneumonitis
  * Grade 3 colitis
Part B1: Number of participants with DLTs | Through Cycle 1 (21 days)
  AEs as per NCI CTCAE version 5.0:
  * Grade 5 not related to disease progression or other causes
  * Grade ≥3 non-hematologic toxicity; exceptions: grade 3 nausea, vomiting or diarrhea controlled in 72 hours; grade 3 fatigue <5 days; grade ≥3 correctable electrolyte abnormalities <72 hours and no clinical complications; grade ≥3 amylase or lipase without clinical pancreatitis
  * Hy's law cases
  * Grade 3 AST or ALT or grade 3 bilirubinemia >5 days
  * Hematologic DLTs:
    * Grade 4 neutropenia or thrombocytopenia >7 days
    * Febrile neutropenia
    * Grade ≥3 thrombocytopenia with bleeding
  * Grade 4 immune-related AEs
  * Grade 3 or 4 non-infectious pneumonitis
  * Grade 3 immune-related AEs, excluding colitis, hepatitis, and pneumonitis, not downgrading to grade ≤2 in 3 days despite maximal supportive care including systemic corticosteroids or to grade 1 or baseline in 14 days
  * Grade 2 pneumonitis not downgrading to grade 1 in 3 days
  * Recurrent grade 2 pneumonitis
  * Grade 3 colitis
Part A: Number of participants with AEs | Day 1 up to approximately 3 years
  Nanrilkefusp alfa related only
Part A1: Number of participants with AEs | Day 1 up to approximately 3 years
  Nanrilkefusp alfa related only
Part B: Number of participants with AEs | Day 1 up to approximately 3 years
  Nanrilkefusp alfa related only
Part B1: Number of participants with AEs | Day 1 up to approximately 3 years
  Nanrilkefusp alfa related only
Part D: Number of participants with AEs | Day 1 up to approximately 3 years
  Nanrilkefusp alfa related only
Part A: Number of participants with serious AEs (SAEs) | Day 1 up to approximately 3 years
  Nanrilkefusp alfa related only
Part A1: Number of participants with SAEs | Day 1 up to approximately 3 years
  Nanrilkefusp alfa related only
Part B: Number of participants with SAEs | Day 1 up to approximately 3 years
  Nanrilkefusp alfa related only
Part B1: Number of participants with SAEs | Day 1 up to approximately 3 years
  Nanrilkefusp alfa related only
Part D: Number of participants with SAEs | Day 1 up to approximately 3 years
  Nanrilkefusp alfa related only
Part A: Number of participants with AEs leading to premature discontinuation of nanrilkefusp alfa | Day 1 up to approximately 3 years
  Nanrilkefusp alfa related only
Part A1: Number of participants with AEs leading to premature discontinuation of nanrilkefusp alfa | Day 1 up to approximately 3 years
  Nanrilkefusp alfa related only
Part B: Number of participants with AEs leading to premature discontinuation of nanrilkefusp alfa | Day 1 up to approximately 3 years
  Nanrilkefusp alfa related only
Part B1: Number of participants with AEs leading to premature discontinuation of nanrilkefusp alfa | Day 1 up to approximately 3 years
  Nanrilkefusp alfa related only
Part D: Number of participants with AEs leading to premature discontinuation of nanrilkefusp alfa | Day 1 up to approximately 3 years
  Nanrilkefusp alfa related only
Part A: Number of participants who died | Day 1 up to approximately 3 years
  Nanrilkefusp alfa-related deaths only
Part A1: Number of participants who died | Day 1 up to approximately 3 years
  Nanrilkefusp alfa-related deaths only
Part B: Number of participants who died | Day 1 up to approximately 3 years
  Nanrilkefusp alfa-related deaths only
Part B1: Number of participants who died | Day 1 up to approximately 3 years
  Nanrilkefusp alfa-related deaths only
Part D: Number of participants who died | Day 1 up to approximately 3 years
  Nanrilkefusp alfa-related deaths only
Part A: Number of participants with nanrilkefusp alfa-related clinical laboratory test abnormalities (coagulation; hematology; clinical chemistry; urinalysis; thyroid and cardiac function) | Day 1 up to approximately 3 years
  The following laboratory parameters will be assessed:
  * Coagulation: Prothrombin time, activated partial thromboplastin time, international normalized ratio, D-dimer, fibrinogen
  * Hematology: Hemoglobin, hematocrit, red blood cell count, reticulocytes, white blood cell count (with full differentiation), absolute lymphocyte count, platelet count
  * Clinical chemistry: Na, K, Cl, phosphate, Mg, Ca, albumin, total protein, ALT, AST, bilirubin (direct, total), alkaline phosphatase, lactate dehydrogenase, creatinine clearance, creatinine, glucose (preferably fasting), urea or blood urea nitrogen, cholesterol, triglyceride, CRP, uric acid, amylase, lipase
  * Urinalysis: pH, glucose, protein, bilirubin, urobilinogen. Microscopic examination: red blood cell count, white blood cell count, epithelial cells, bacteria
  * Thyroid function: TSH, free triiodothyronine (T3), free thyroxine (T4)
  * Cardiac function: Cardiac troponin T
Part A1: Number of participants with nanrilkefusp alfa-related clinical laboratory test abnormalities (coagulation; hematology; clinical chemistry; urinalysis; thyroid and cardiac function) | Day 1 up to approximately 3 years
  The following laboratory parameters will be assessed:
  * Coagulation: Prothrombin time, activated partial thromboplastin time, international normalized ratio, D-dimer, fibrinogen
  * Hematology: Hemoglobin, hematocrit, red blood cell count, reticulocytes, white blood cell count (with full differentiation), absolute lymphocyte count, platelet count
  * Clinical chemistry: Na, K, Cl, phosphate, Mg, Ca, albumin, total protein, ALT, AST, bilirubin (direct, total), alkaline phosphatase, lactate dehydrogenase, creatinine clearance, creatinine, glucose (preferably fasting), urea or blood urea nitrogen, cholesterol, triglyceride, CRP, uric acid, amylase, lipase
  * Urinalysis: pH, glucose, protein, bilirubin, urobilinogen. Microscopic examination: red blood cell count, white blood cell count, epithelial cells, bacteria
  * Thyroid function: TSH, free triiodothyronine (T3), free thyroxine (T4)
  * Cardiac function: Cardiac troponin T
Part B: Number of participants with nanrilkefusp alfa-related clinical laboratory test abnormalities (coagulation; hematology; clinical chemistry; urinalysis; thyroid and cardiac function) | Day 1 up to approximately 3 years
  The following laboratory parameters will be assessed:
  * Coagulation: Prothrombin time, activated partial thromboplastin time, international normalized ratio, D-dimer, fibrinogen
  * Hematology: Hemoglobin, hematocrit, red blood cell count, reticulocytes, white blood cell count (with full differentiation), absolute lymphocyte count, platelet count
  * Clinical chemistry: Na, K, Cl, phosphate, Mg, Ca, albumin, total protein, ALT, AST, bilirubin (direct, total), alkaline phosphatase, lactate dehydrogenase, creatinine clearance, creatinine, glucose (preferably fasting), urea or blood urea nitrogen, cholesterol, triglyceride, CRP, uric acid, amylase, lipase
  * Urinalysis: pH, glucose, protein, bilirubin, urobilinogen. Microscopic examination: red blood cell count, white blood cell count, epithelial cells, bacteria
  * Thyroid function: TSH, free triiodothyronine (T3), free thyroxine (T4)
  * Cardiac function: Cardiac troponin T
Part B1: Number of participants with nanrilkefusp alfa-related clinical laboratory test abnormalities (coagulation; hematology; clinical chemistry; urinalysis; thyroid and cardiac function) | Day 1 up to approximately 3 years
  The following laboratory parameters will be assessed:
  * Coagulation: Prothrombin time, activated partial thromboplastin time, international normalized ratio, D-dimer, fibrinogen
  * Hematology: Hemoglobin, hematocrit, red blood cell count, reticulocytes, white blood cell count (with full differentiation), absolute lymphocyte count, platelet count
  * Clinical chemistry: Na, K, Cl, phosphate, Mg, Ca, albumin, total protein, ALT, AST, bilirubin (direct, total), alkaline phosphatase, lactate dehydrogenase, creatinine clearance, creatinine, glucose (preferably fasting), urea or blood urea nitrogen, cholesterol, triglyceride, CRP, uric acid, amylase, lipase
  * Urinalysis: pH, glucose, protein, bilirubin, urobilinogen. Microscopic examination: red blood cell count, white blood cell count, epithelial cells, bacteria
  * Thyroid function: TSH, free triiodothyronine (T3), free thyroxine (T4)
  * Cardiac function: Cardiac troponin T
Part D: Number of participants with nanrilkefusp alfa-related clinical laboratory test abnormalities (coagulation; hematology; clinical chemistry; urinalysis; thyroid and cardiac function) | Day 1 up to approximately 3 years
  The following laboratory parameters will be assessed:
  * Coagulation: Prothrombin time, activated partial thromboplastin time, international normalized ratio, D-dimer, fibrinogen
  * Hematology: Hemoglobin, hematocrit, red blood cell count, reticulocytes, white blood cell count (with full differentiation), absolute lymphocyte count, platelet count
  * Clinical chemistry: Na, K, Cl, phosphate, Mg, Ca, albumin, total protein, ALT, AST, bilirubin (direct, total), alkaline phosphatase, lactate dehydrogenase, creatinine clearance, creatinine, glucose (preferably fasting), urea or blood urea nitrogen, cholesterol, triglyceride, CRP, uric acid, amylase, lipase
  * Urinalysis: pH, glucose, protein, bilirubin, urobilinogen. Microscopic examination: red blood cell count, white blood cell count, epithelial cells, bacteria
  * Thyroid function: TSH, free triiodothyronine (T3), free thyroxine (T4)
  * Cardiac function: Cardiac troponin T

SECONDARY OUTCOMES:
Part A: Nanrilkefusp alfa concentration profile, Cycle 1 Day 1, 1 hour (+/-15 minutes) | Cycle 1 Day 1, 1 hour (+/-15 minutes)
  After 12 μg/kg nanrilkefusp alfa administration
Part A1: Nanrilkefusp alfa concentration profile, Cycle 1 Day 1, 1 hour (+/-15 minutes) | Cycle 1 Day 1, 1 hour (+/-15 minutes)
  After 12 μg/kg nanrilkefusp alfa administration
Part B: Nanrilkefusp alfa concentration profile, Cycle 1 Day 1, 1 hour (+/-15 minutes) | Cycle 1 Day 1, 1 hour (+/-15 minutes)
  After 12 μg/kg nanrilkefusp alfa administration
Part D: Nanrilkefusp alfa concentration profile, Cycle 1 Day 1, 1 hour (+/-15 minutes) | Cycle 1 Day 1, 1 hour (+/-15 minutes)
  After 12 μg/kg nanrilkefusp alfa administration
Part A: Nanrilkefusp alfa concentration profile, Cycle 1 Day 1, 4 hours (+/-15 minutes) | Cycle 1 Day 1, 4 hours (+/-15 minutes)
  After 12 μg/kg nanrilkefusp alfa administration
Part A1: Nanrilkefusp alfa concentration profile, Cycle 1 Day 1, 4 hours (+/-15 minutes) | Cycle 1 Day 1, 4 hours (+/-15 minutes)
  After 12 μg/kg nanrilkefusp alfa administration
Part B: Nanrilkefusp alfa concentration profile, Cycle 1 Day 1, 4 hours (+/-15 minutes) | Cycle 1 Day 1, 4 hours (+/-15 minutes)
  After 12 μg/kg nanrilkefusp alfa administration
Part D: Nanrilkefusp alfa concentration profile, Cycle 1 Day 1, 4 hours (+/-15 minutes) | Cycle 1 Day 1, 4 hours (+/-15 minutes)
  After 12 μg/kg nanrilkefusp alfa administration
Part A: Overall activation levels of Ki-67+ CD8+ T cells on day 6 of cycle 1 | Day 6 of Cycle 1
  At 12 μg/kg nanrilkefusp alfa
Part A1: Overall activation levels of Ki-67+ CD8+ T cells on day 6 of cycle 1 | Day 6 of Cycle 1
  At 12 μg/kg nanrilkefusp alfa
Part B: Overall activation levels of Ki-67+ CD8+ T cells on day 6 of cycle 1 | Day 6 of Cycle 1
  At 12 μg/kg nanrilkefusp alfa
Part D: Overall activation levels of Ki-67+ CD8+ T cells on day 6 of cycle 1 | Day 6 of Cycle 1
  At 12 μg/kg nanrilkefusp alfa
Part A: Overall activation levels of Ki-67+ CD8+ CD45RO+ CD45RA- T cells on day 6 of cycle 1 | Day 6 of Cycle 1
  At 12 μg/kg nanrilkefusp alfa
Part A1: Overall activation levels of Ki-67+ CD8+ CD45RO+ CD45RA- T cells on day 6 of cycle 1 | Day 6 of Cycle 1
  At 12 μg/kg nanrilkefusp alfa
Part B: Overall activation levels of Ki-67+ CD8+ CD45RO+ CD45RA- T cells on day 6 of cycle 1 | Day 6 of Cycle 1
  At 12 μg/kg nanrilkefusp alfa
Part D: Overall activation levels of Ki-67+ CD8+ CD45RO+ CD45RA- T cells on day 6 of cycle 1 | Day 6 of Cycle 1
  At 12 μg/kg nanrilkefusp alfa
Part A: Overall activation levels of Ki-67+ CD4+ T cells on day 6 of cycle 1 at 12 μg/kg nanrilkefusp alfa | Day 6 of Cycle 1
  At 12 μg/kg nanrilkefusp alfa
Part A1: Overall activation levels of Ki-67+ CD4+ T cells on day 6 of cycle 1 at 12 μg/kg nanrilkefusp alfa | Day 6 of Cycle 1
  At 12 μg/kg nanrilkefusp alfa
Part B: Overall activation levels of Ki-67+ CD4+ T cells on day 6 of cycle 1 at 12 μg/kg nanrilkefusp alfa | Day 6 of Cycle 1
  At 12 μg/kg nanrilkefusp alfa
Part D: Overall activation levels of Ki-67+ CD4+ T cells on day 6 of cycle 1 at 12 μg/kg nanrilkefusp alfa | Day 6 of Cycle 1
  At 12 μg/kg nanrilkefusp alfa
Part A: Overall activation levels of Ki-67+ NK cells on day 6 of cycle 1 at 12 μg/kg nanrilkefusp alfa | Day 6 of Cycle 1
  At 12 μg/kg nanrilkefusp alfa
Part A1: Overall activation levels of Ki-67+ NK cells on day 6 of cycle 1 at 12 μg/kg nanrilkefusp alfa | Day 6 of Cycle 1
  At 12 μg/kg nanrilkefusp alfa
Part B: Overall activation levels of Ki-67+ NK cells on day 6 of cycle 1 at 12 μg/kg nanrilkefusp alfa | Day 6 of Cycle 1
  At 12 μg/kg nanrilkefusp alfa
Part D: Overall activation levels of Ki-67+ NK cells on day 6 of cycle 1 at 12 μg/kg nanrilkefusp alfa | Day 6 of Cycle 1
  At 12 μg/kg nanrilkefusp alfa
Part A: Overall activation levels of Ki-67+ NKT cells on day 6 of cycle 1 at 12 μg/kg nanrilkefusp alfa | Day 6 of Cycle 1
  At 12 μg/kg nanrilkefusp alfa
Part A1: Overall activation levels of Ki-67+ NKT cells on day 6 of cycle 1 at 12 μg/kg nanrilkefusp alfa | Day 6 of Cycle 1
  At 12 μg/kg nanrilkefusp alfa
Part B: Overall activation levels of Ki-67+ NKT cells on day 6 of cycle 1 at 12 μg/kg nanrilkefusp alfa | Day 6 of Cycle 1
  At 12 μg/kg nanrilkefusp alfa
Part D: Overall activation levels of Ki-67+ NKT cells on day 6 of cycle 1 at 12 μg/kg nanrilkefusp alfa | Day 6 of Cycle 1
  At 12 μg/kg nanrilkefusp alfa
Part A: Overall activation levels of Ki-67+ Treg cells on day 6 of cycle 1 at 12 μg/kg nanrilkefusp alfa | Day 6 of Cycle 1
  At 12 μg/kg nanrilkefusp alfa
Part A1: Overall activation levels of Ki-67+ Treg cells on day 6 of cycle 1 at 12 μg/kg nanrilkefusp alfa | Day 6 of Cycle 1
  At 12 μg/kg nanrilkefusp alfa
Part B: Overall activation levels of Ki-67+ Treg cells on day 6 of cycle 1 at 12 μg/kg nanrilkefusp alfa | Day 6 of Cycle 1
  At 12 μg/kg nanrilkefusp alfa
Part D: Overall activation levels of Ki-67+ Treg cells on day 6 of cycle 1 at 12 μg/kg nanrilkefusp alfa | Day 6 of Cycle 1
  At 12 μg/kg nanrilkefusp alfa
Part A: Objective response rate (ORR) | Day 1 up to approximately 3 years
  Based on investigator review of radiographic images according to Response Evaluation Criteria In Solid Tumors for immune-based therapeutics (iRECIST)
Part A1: ORR | Day 1 up to approximately 3 years
  Based on investigator review of radiographic images according to iRECIST
Part B: ORR | Day 1 up to approximately 3 years
  Based on investigator review of radiographic images according to iRECIST
Part D: ORR | Day 1 up to approximately 3 years
  Based on investigator review of radiographic images according to iRECIST
Part A: Duration of response (DoR) | Day 1 up to approximately 3 years
  DoR according to iRECIST
Part A1: DoR | Day 1 up to approximately 3 years
  DoR according to iRECIST
Part B: DoR | Day 1 up to approximately 3 years
  DoR according to iRECIST
Part D: DoR | Day 1 up to approximately 3 years
  DoR according to iRECIST
Part A: Clinical benefit rate (CBR) | Day 1 up to approximately 3 years
  CBR according to iRECIST
Part A1: CBR | Day 1 up to approximately 3 years
  CBR according to iRECIST
Part B: CBR | Day 1 up to approximately 3 years
  CBR according to iRECIST
Part D: CBR | Day 1 up to approximately 3 years
  CBR according to iRECIST
Part A: Progression-free survival (PFS) | Day 1 up to approximately 3 years
  PFS according to iRECIST
Part A1: PFS | Day 1 up to approximately 3 years
  PFS according to iRECIST
Part B: PFS | Day 1 up to approximately 3 years
  PFS according to iRECIST
Part D: PFS | Day 1 up to approximately 3 years
  PFS according to iRECIST
Part A: Number of participants with anti-drug antibodies (ADAs) at the end of treatment | End of treatment with nanrilkefusp alfa
  Against nanrilkefusp alfa
Part A1: Number of participants with ADAs at the end of treatment | End of treatment with nanrilkefusp alfa
  Against nanrilkefusp alfa
Part B: Number of participants with ADAs at the end of treatment | End of treatment with nanrilkefusp alfa
  Against nanrilkefusp alfa
Part B1: Number of participants with ADAs at the end of treatment | End of treatment with nanrilkefusp alfa
  Against nanrilkefusp alfa
Part D: Number of participants with ADAs at the end of treatment | End of treatment with nanrilkefusp alfa
  Against nanrilkefusp alfa

CONTACTS AND LOCATIONS:
Overall Officials: Stephane Champiat, Dr., Principal Investigator — Institute Gustave Roussy, Villejuif, France
Locations (12):
- United States (3):
  - Yale Cancer Center, New Haven, Connecticut
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
- Masarykův Onkologický Ústav Brno Klinika komplexní onkologické péče, Brno, Czechia
- France (6):
  - Centre Léon Bérard, Lyon
  - Hôpitaux Universitaires de Marseille Timone, Marseille
  - Hopital Saint Louis, Paris
  - Institut Gustave Roussy, Paris
  - Institut de Cancerologie de L'Ouest, Saint-Herblain
  - Institut Claudius Regaud, Toulouse
- Spain (2):
  - Vall d'Hebron Institute of Oncology, Barcelona
  - University Hospital Sanchinarro, Madrid

IPD SHARING:
Plan to Share IPD: No